CLINICAL TRIAL: NCT02552290
Title: Effects of Cervicothoracic Manipulation and Passive Stretching to the Upper Trapezius Muscle on Pressure Pain Thresholds and Cervical Range of Motion on Healthy Individuals
Brief Title: Immediate Effects Cervicothoracic Manipulation Versus Passive Upper Trapezius Stretch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Emilio J Puentedura, PT, DPT, PhD, Associate Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1303-4412
Record Dates: First submitted 2015-09-14; First posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cervicothoracic manipulation (Active Comparator): Description of a Right C7/T1 manipulation. The subject will lie prone. The therapist will stand on the L side of the subject facing in a cephalic direction (towards the patient's head). The therapist's right hand makes contact with the thumb on the right side of the spinous process of the first thoracic vertebra. The therapist left hand supports the head making contact on the temporal bone. The hand/neck is gently laterally flexed to the right, until slight tension is palpated in the tissues. A high-velocity low-amplitude thrust will be applied towards the subjects left side. If cavitation does not occur (an audible pop) the subject will be repositioned and the manipulation attempted a second time. A maximum of 2 attempts will be performed for each side of the neck.
  Interventions: Other: Cervicothoracic manipulation
- Upper trapezius stretch (Active Comparator): The subjects will be in a supine position. A researcher will passively place the subject's head into flexion, side-bending away and rotation towards the side to be stretched until the muscle barrier is met. The researcher will depress the subject's shoulder with 100 Newtons of force measured with a Micro FET pressure dynamometer (Hoggan Health Industries, Salt Lake City, UT).) Once this pressure amount is achieved the stretch will be held for 30 seconds. This will be repeated two times on each side.
  The subject will be asked to provide continuous feedback about the stretch felt and the degree of discomfort (if any) felt during the 30 second stretches.
  Interventions: Other: Upper Trapezius Stretch
- Control group (Other): Subjects assigned to the control group will receive no intervention. They will stay behind the curtained research area for approximately 3 minutes in a seated position.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Upper Trapezius Stretch — Sustained stretch of upper trapezius muscle
  Arms: Upper trapezius stretch
Other: Cervicothoracic manipulation — Manipulation to the cervicothoracic spine
  Arms: Cervicothoracic manipulation
Other: No intervention — Wait
  Arms: Control group

SUMMARY:
The proposed project seeks to evaluate the influence of cervicothoracic (CT) manipulation and passive stretching to the upper trapezius on pressure pain thresholds and range of motion (ROM) in individuals without recent complain of neck pain.

DETAILED DESCRIPTION:
Not needed

ELIGIBILITY:
Inclusion Criteria:

1. No current history or past history of neck pain; able to lie on back or stomach without difficulty

Exclusion Criteria:

1. 'Red flag' items indicated in your Neck Medical Screening Questionnaire such as history of a tumor, bone fracture, metabolic diseases, Rheumatoid Arthritis, osteoporosis, severe atherosclerosis, prolonged history of steroid use, etc.
2. History of neck whiplash injury
3. Diagnosis from your physician of cervical spinal stenosis (narrowing of spinal canal) or presence of symptoms (pain, pins and needles, numbness) down both arms
4. Presence of central nervous system involvement such as exaggerated reflexes, changes in sensation in the hands, muscle wasting in the hands, impaired sensation of the face, altered taste, and presence of abnormal reflexes
5. Evidence of neurological signs consistent with nerve root entrapment (pinched nerve in the neck)
6. Prior surgery to your neck or upper back
7. A medical condition which may influence assessment of pain or pressure pain thresholds (i.e. taking analgesics, sedatives, history of substance abuse, or cognitive deficiency)
8. Diagnosis from your physician of fibromyalgia syndrome
9. Currently pregnant, or could be pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Cervical Range of Motion | Immediately after the intervention
  Cervical Range of Motion in each cardinal plane (sagittal, coronal and transverse) will be measured in angular degrees using a CROM device

SECONDARY OUTCOMES:
Pain Pressure Threshold | Two minutes and 5 Minutes after the intervention
  Pain Pressure Threshold measured using a standard handheld algometer with 1 cm round tip

CONTACTS AND LOCATIONS:
Overall Officials: Emilio J Puentedura, PT, DPT, PhD, Principal Investigator — UNLV
Locations (1):
- University of Nevada Las Vegas - Department of Physical Therapy, Las Vegas, Nevada, United States